CLINICAL TRIAL: NCT05618938
Title: Effects of Rocabado's Approach Versus Kraus Exercise Therapy on Pain and Disability in Patients With Temporomandibular Dysfunction
Brief Title: Effects of Rocabado's Approach Versus Kraus Exercise Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0151 Amna
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Temporomandibular Dysfunction
Keywords: Rocabado's Approach; Kraus exercises; Disability
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group: A Rocabado's approach (Experimental): 1. Rest position of the tongue: The anterior 1/3 of the tongue is placed at the palate with mild pressure.
  2. Control of TMJ rotation: The jaw is repeatedly opened and closed with the anterior 1/3 of the tongue on the palate.
  3. Rhythmic stabilization technique: Gentle isometrics in the resting position are performed for jaw opening, closing, and lateral deviation.
  4. Axial extension of the neck: Combined upper cervical flexion with lower cervical extension.
  Interventions: Other: Rocabado's approach
- Group B: Kraus exercises (Experimental): Group B will be treated with Kraus exercises. Kraus exercises will be comprised of eight exercise programs.
  1. Tongue position at rest: The patient will be instructed to maintain a resting tongue position except during function, which involves the tip of the tongue sitting on the palate with the tip resting just posterior to the upper incisors
  2. Teeth apart: the patient will be educated to maintain the teeth apart can be therapeutic, which facilitates the resting tongue position
  3. Nasal-diaphragmatic breathing: The patient will be instructed in nasal breathing to facilitate function of the diaphragm, which reinforces positioning of both the tongue and teeth
  4. Tongue up and wiggle: Place the tongue to the palate, then move the jaw from side to side.
  5. Strengthening: Resisted closing via self-manual resistance using tongue depressor between lower incisors: 5-10-second contractions.
  Interventions: Other: Kraus exercises

INTERVENTIONS:
Other: Rocabado's approach — Group A will be treated with Rocabado's approach. Rocabado' approach will be comprised of six exercises.
  1. Rest position of the tongue
  2. Control of TMJ rotation
  3. Rhythmic stabilization technique
  4. Axial extension of the neck The patients will receive Rocabado's approach consisting 6 repetitions six times a day thrice per week for four weeks
  Arms: Group: A Rocabado's approach
Other: Kraus exercises — Group B will be treated with Kraus exercises. Kraus exercises will be comprised of eight exercise programs.
  1. Tongue position at rest
  2. Teeth apart: the patient will be educated to maintain the teeth apart can be therapeutic, which facilitates the resting tongue position
  3. Nasal-diaphragmatic breathing
  4. Tongue up and wiggle
  5. Strengthening
  6. Touch and bite: Proprioceptive re-education: Lateral deviation The patients will receive Kraus exercises with the frequency of 2 sets and 10 repetitions twice a day three times per week for four weeks
  Arms: Group B: Kraus exercises

SUMMARY:
TMJ dysfunction is linked to trauma, joint overloading owing to para-functional behaviors, mechanical stress, and metabolic issues. Myofascial pain and dysfunction, functional derangement, and osteoarthrosis are the three most frequent TMJ-related disorders. Temporomandibular joint disorders are a type of craniofacial problems. They affect the temporomandibular joint, muscles of mastication, and other musculoskeletal tissues. The most common clinical sign and symptoms associated with TMJ dysfunction are orofacial pain and clicking. The aim of study will be to compare the effects of Rocabado's approach versus Kraus therapy on Pain and Disability in patients with temporomandibular dysfunction.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at FMH Physiotherapy Clinic and Boston Physiotherapy Clinic Lahore through consecutive sampling technique on 40 patients which will be allocated using random sampling through opaque sealed enveloped into Group A and Group B. Group A will be treated with Rocabado's approach and Group B will be treated with Kraus exercises. Outcome measures tools will be conducted through NPRS, TMD disability index, Fonseca questionnaire after four weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between the ages of 30 to 60 years
* Patients with jaw pain
* Patients with limited jaw range of motion and associated joint pain
* Patients with TMJ clicking sounds
* Patients with pain upon muscle and joint palpation

Exclusion Criteria:

* Diagnosis of ear, nose, and throat medical pathology underlying the tinnitus;
* Neurological problems that could potentially cause the tinnitus
* Inability to read, understand, and complete the questionnaires or understand and follow commands (e.g., illiteracy, dementia, or blindness)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-02-04 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.
  pre and post followup on 4th week
Temporomandibular Joint Disability Index Questionnaire: | 4th week
  The TMD Disability Index is a ten-question questionnaire that is based on the Oswestry Back Pain Questionnaire and the Neck Pain and Disability Questionnaire. 12 It is TMJ-specific, comprising specialized TMJ tasks (instrument playing, speech, dental care, and so on); it delivers a score ranging from 20 to 100.
  pre and post followup on 4th week
Fonseca's Questionnaire for severity | 4th week
  TMD diseases are classified using the Fonseca questionnaire into mild, moderate, severe, or no disease. It consists of ten questions about temporomandibular joint pain, head, back, and chewing discomfort, parafunctional habits, movement limits, joint clicking, perception of malocclusion, and emotional stress sensation.
  pre and post followup on 4th week

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Fatima Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scrivani SJ, Khawaja SN, Bavia PF. Nonsurgical Management of Pediatric Temporomandibular Joint Dysfunction. Oral Maxillofac Surg Clin North Am. 2018 Feb;30(1):35-45. doi: 10.1016/j.coms.2017.08.001. PMID 29153236
- [Background] Matsubara R, Yanagi Y, Oki K, Hisatomi M, Santos KC, Bamgbose BO, Fujita M, Okada S, Minagi S, Asaumi J. Assessment of MRI findings and clinical symptoms in patients with temporomandibular joint disorders. Dentomaxillofac Radiol. 2018 May;47(4):20170412. doi: 10.1259/dmfr.20170412. Epub 2018 Feb 22. PMID 29451403
- [Background] Dimitroulis G. Temporomandibular joint surgery: what does it mean to the dental practitioner? Aust Dent J. 2011 Sep;56(3):257-64. doi: 10.1111/j.1834-7819.2011.01351.x. PMID 21884140
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Slade GD, Bair E, Greenspan JD, Dubner R, Fillingim RB, Diatchenko L, Maixner W, Knott C, Ohrbach R. Signs and symptoms of first-onset TMD and sociodemographic predictors of its development: the OPPERA prospective cohort study. J Pain. 2013 Dec;14(12 Suppl):T20-32.e1-3. doi: 10.1016/j.jpain.2013.07.014. PMID 24275221
- [Background] Yadav S, Yang Y, Dutra EH, Robinson JL, Wadhwa S. Temporomandibular Joint Disorders in Older Adults. J Am Geriatr Soc. 2018 Jul;66(6):1213-1217. doi: 10.1111/jgs.15354. Epub 2018 May 2. PMID 29719041
- [Background] Lora VR, Canales Gde L, Goncalves LM, Meloto CB, Barbosa CM. Prevalence of temporomandibular disorders in postmenopausal women and relationship with pain and HRT. Braz Oral Res. 2016 Aug 22;30(1):e100. doi: 10.1590/1807-3107BOR-2016.vol30.0100. PMID 27556676
- [Background] Ernst M, Schenkenberger AE, Domin M, Kordass B, Lotze M. Effects of centric mandibular splint therapy on orofacial pain and cerebral activation patterns. Clin Oral Investig. 2020 Jun;24(6):2005-2013. doi: 10.1007/s00784-019-03064-y. Epub 2019 Sep 13. PMID 31520181
- [Background] Seifi M, Ebadifar A, Kabiri S, Badiee MR, Abdolazimi Z, Amdjadi P. Comparative effectiveness of Low Level Laser therapy and Transcutaneous Electric Nerve Stimulation on Temporomandibular Joint Disorders. J Lasers Med Sci. 2017 Summer;8(Suppl 1):S27-S31. doi: 10.15171/jlms.2017.s6. Epub 2017 Aug 29. PMID 29071032
- [Background] Lopez-Martos R, Gonzalez-Perez LM, Ruiz-Canela-Mendez P, Urresti-Lopez FJ, Gutierrez-Perez JL, Infante-Cossio P. Randomized, double-blind study comparing percutaneous electrolysis and dry needling for the management of temporomandibular myofascial pain. Med Oral Patol Oral Cir Bucal. 2018 Jul 1;23(4):e454-e462. doi: 10.4317/medoral.22488. PMID 29924769